CLINICAL TRIAL: NCT07226765
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Maridebart Cafraglutide in Adult Participants With Obstructive Sleep Apnea Not on Positive Airway Pressure Therapy and Living With Overweight or Obesity (MARITIME-OSA-2)
Brief Title: Maridebart Cafraglutide Versus Placebo in Adult Participants With Obstructive Sleep Apnea Not on Positive Airway Pressure (PAP) Therapy
Acronym: MARITIME-OSA-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20250002
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; OSA; Overweight; Obesity; Maridebart Cafraglutide; AMG 133; MariTide
MeSH Terms: conditions — Sleep Apnea, Obstructive; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maridebart Cafraglutide (Experimental): Participants will receive maridebart cafraglutide subcutaneously (SC).
  Interventions: Drug: Maridebart cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart cafraglutide — Participants will receive maridebart cafraglutide SC.
  Other Names: AMG 133; MariTide
  Arms: Maridebart Cafraglutide
Drug: Placebo — Participants will receive placebo SC.
  Arms: Placebo

SUMMARY:
This Phase 3 clinical trial is designed to evaluate the efficacy and safety of maridebart cafraglutide compared to placebo over a 52-week period in adults with obstructive sleep apnea (OSA) who are not on PAP therapy and are living with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an AHI of 15 or higher on polysomnography (PSG) at Day 1 before randomization.
* Body Mass Index (BMI) of 27 kg/m^2 or more at the time of screening.
* History of at least one unsuccessful attempt at weight loss through diet and exercise.
* Participants must not have used PAP therapy for at least 4 weeks before screening, are unwilling/unable to use PAP, and do not plan to use PAP therapy during the study.

Exclusion Criteria:

* Individuals who have had any previous or planned upper airway surgery for sleep apnea or major ear, nose, or throat surgery.
* Those with significant craniofacial abnormalities that may affect breathing at screening.
* Participants diagnosed with Central Apnea with a percentage of central apneas/hypopneas of 50% or more, or those diagnosed with Cheyne Stokes Respiration.
* Active device treatment of OSA (eg, PAP, oral appliances), or other treatments, that in the opinion of the investigator, may interfere with study outcomes, unless willing to stop treatment at screening and throughout the study.
* Individuals with respiratory diseases like obesity hypoventilation syndrome or daytime hypercapnia, neuromuscular diseases or other conditions that could interfere with the trial results, according to the investigator's opinion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2028-09-13 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea-hypopnea Index (AHI) from baseline at Week 52 | At Week 52

SECONDARY OUTCOMES:
Percent Change in AHI from baseline at Week 52 | At Week 52
Participants Achieving ≥ 50% AHI Reduction from baseline at Week 52 | At Week 52
Participants Achieving AHI < 5 or AHI 5 to 14 with Epworth Sleepiness Scale (ESS) ≤ 10 from baseline at Week 52 | At Week 52
Percent Change in Body Weight from baseline at Week 52 | At Week 52
Change in Sleep Apnea-specific Hypoxic Burden (SASHB) from baseline at Week 52 | At Week 52
Change in High Sensitivity C-reactive Protein (hs-CRP) from baseline at Week 52 | At Week 52
Change in Systolic Blood Pressure (SBP) from baseline at Week 48 | At Week 48
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Sleep-related Impairment 8a Score from baseline at Week 52 | At Week 52

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (11):
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Teradan Clinical Trials, Brandon, Florida
  - Destiny Research Center, Palmetto Bay, Florida
  - Clinical Research Center Of Florida, Pompano Beach, Florida
  - Basil Clinical, Laurelton, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - FutureSearch Trials of Neurology, Austin, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Australia (2):
  - Woolcock Institute of Medical Research, Macquarie Park, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
- Canada (2):
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Wharton Medical Clinic, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com